CLINICAL TRIAL: NCT06046456
Title: Prenatal Affective Cognitive Training to Reduce the Risk of Postpartum Depression (PACT): Study Protocol for a Randomized Controlled Trial
Brief Title: Prenatal Affective Cognitive Training to Reduce the Risk of Postpartum Depression (PACT)
Acronym: PACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R7-A182
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-08

CONDITIONS: Postpartum Depression; Emotional Regulation; Cognitive Function 1, Social; Pregnancy Related; Mother-Child Relations
MeSH Terms: conditions — Depression, Postpartum; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACT (Experimental): Receive the intervention
  Interventions: Other: Prenatal Affective CogntiiveTraining
- CAU (No Intervention): Receive care as usual, i.e., the standard care provided to pregnant women without any additional experimental interventions. It typically involves routine prenatal care, which may include regular check-ups, medical assessments, and general support from healthcare professionals

INTERVENTIONS:
Other: Prenatal Affective CogntiiveTraining — A psychological intervention using computer- and virtual reality based exercises to modify negative cognitive bias and improve emotion regulation
  Arms: PACT

SUMMARY:
Many pregnant women face the risk of experiencing depression after giving birth, especially if they've previously dealt with depression.

The goal of this study, is to test if our newly developed Prenatal Affective Cognitive Training (PACT) intervention, can decrease the likelihood of post partum depression. In the study, 226 pregnant women, some of whom are considered high risk due to past mental illness or psycho-social risk factors, will participate. The high-risk women will be divided into two groups. One group will undergo the PACT training, which involves computer and virtual reality exercises spanning five weeks, designed to improve mood and emotional regulation. The other group will receive usual care. The study also involves a low-risk group (n=146), although these individuals are not part of the intervention trial but are merely followed up with the same assessments for background comparisons.The main aim is to observe whether the women who undergo PACT intervention are less prone to depression after childbirth compared to those who do not.

This study has potential to offer a simple, non-invasive method to bolster mental health in expectant mothers, which could also positively impact their infants.

ELIGIBILITY:
Inclusion Criteria for General Pregnant Population:

* Second or third trimester pregnancy.
* Age ≥ 18 years.
* Ability to speak and read Danish.

Inclusion Criteria for High-Risk Pregnant Group:

* Either:
* Negative cognitive bias in emotional reactivity to infant distress (cut-off > 96 on a scale from 0-100).
* High-risk status according to the Antenatal Risk Questionnaire (ANRQ) which means:
* Personal history of severe mental illness.
* Experienced childhood emotional, physical, or sexual abuse.
* Total score on psycho-social risk factors is above the cut-off (> 23).

Inclusion Criteria for Low-Risk Pregnant Group:

* Absence of a personal or family history of mental illness.
* Absence of negative bias.
* Three or fewer of the additional risk factors mentioned above.

General Exclusion Criteria:

* Schizophrenia.
* Current substance use disorder.
* Score of 9 or more on the Hamilton Depression Rating Scale-6 items (HDRS-6), indicating moderate depression.
* Pregnant women diagnosed with a personality disorder (note: they will still be included at baseline and follow-up after birth but will be excluded from randomization).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of PPD during the first six months after birth, assessed with the Present State Examination (PSE), which is a part of Schedules for Clinical Assessment in Neuropsychiatry (SCAN) | Six months after birth
  The primary outcome is the difference between mothers receiving PACT versus CAU in the incidence of PPD during the first six months after birth, assessed by a clinician blind to group status with the Present State Examination (PSE), which is a part of Schedules for Clinical Assessment in Neuropsychiatry (SCAN)

SECONDARY OUTCOMES:
Change in negative cognitive bias | In third trimester of pregnancy
  Differences between participants receiving PACT and CAU in the change in negatively biased cognitive processing of infant stimuli from baseline to follow-up during pregnancy (T1) as measured with computerized testing
Self-rated depressive symptoms | Within six weeks after birth
  Differences between participants receiving PACT and CAU in severity of depressive symptoms during the first six weeks after birth measured with the Edinburgh Postpartum Depression Scale
Self-rated parental stress | Six months after birth
  Self-rated parental stress with the Parental Stress Scale at six months after birth.

OTHER OUTCOMES:
Infant development | Eight - eighteen months after birth
  Tertiary outcome involve assessing differences in infant development as measured with the Bayley Scales version 4 between the PACT and CAU groups
Mother-child interaction | Eight - eighteen months after birth
  Tertiary outcome involve assessing differences in mother-child interaction measures (e.g., sensitivity, intrusiveness, dyadic reciprocity and neural synchrony) between the PACT and CAU groups as measured with behavioural coding (Coding Interactive Behaviour) and fNIRS brain scan.
Change in affective cognition | Third trimester of pregnancy
  Tertiary outcome involve assessing differences in the changes in facial expressions and visual attention towards infant stimuli (from T0 to T1 during pregnancy) between the PACT and CAU groups, as measured with computerized testing

CONTACTS AND LOCATIONS:
Overall Officials: Kamill W Miskowiak, DMsc, Principal Investigator — Mental Health Services in the Capital Region of Denmark
Locations (1):
- Mental Health Services in The Capital Region of Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjertrup AJ, Kofoed J, Egmose I, Wendelboe K, Southgate V, Vaever MS, Miskowiak KW. Prenatal affective cognitive training to reduce the risk of postpartum depression (PACT): study protocol for a randomized controlled trial. Trials. 2024 Jul 15;25(1):478. doi: 10.1186/s13063-024-08316-1. PMID 39010232